CLINICAL TRIAL: NCT07020845
Title: An Investigation on Artificial Intelligence Literacy and E-Health Literacy of Patients With Fibromyalgia Syndrome
Brief Title: Artificial Intelligence, and E-Health Literacy in Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Gulseren Demir Karakilic (Other)
Responsible Party: Sponsor-Investigator, Gulseren Demir Karakilic, Assistant Professor, Principal Investigator, Bozok University
Organization: Bozok University (Other)
Other Study IDs: 2024-GOKAEK-2411_2024.10.16_16
Record Dates: First submitted 2025-06-03; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Fibromyalgia Syndrome; Healthy Controls Group - Age and Sex-matched
Keywords: Fibromyalgia Syndrome; Artificial Intelligence Literacy; Electronic Health Literacy; Revised Fibromyalgia Impact Questionnaire; Beck Depression Inventory; Beck Anxiety Inventory
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the patient group: Patients aged 18 to 50 who attended the Physical Medicine and Rehabilitation outpatient clinic at Bozok University Faculty of Medicine, met the 2016 American College of Rheumatology fibromyalgia diagnostic criteria, demonstrated adequate cognitive function, were literate, and consented to participate were enrolled as the patient group
  Interventions: Other: Observation only
- The control group: The control group consisted of healthy volunteers matched to the patient group in terms of age and sex, aged 18-50 years, with intact cognitive function and literacy skills, no reported health issues, and who willingly consented to participate in the study
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only — This is an observational study with no intervention applied to participants. Data were collected through questionnaires and clinical assessments only

SUMMARY:
This cross-sectional observational study aimed to assess electronic health literacy and artificial intelligence literacy among individuals diagnosed with fibromyalgia syndrome, with particular focus on artificial intelligence literacy. Although general health literacy has been investigated in this patient population, digital and artificial intelligence-related competencies have not been sufficiently studied. The research included 106 individuals diagnosed with fibromyalgia syndrome and 106 age- and sex-matched healthy volunteers, recruited between December 2024 and May 2025. All participants completed a series of standardized questionnaires, including the Revised Fibromyalgia Impact Questionnaire, the Beck Depression Inventory, the Beck Anxiety Inventory, the Electronic Health Literacy Scale, and the Artificial Intelligence Literacy Scale. The study explored demographic, clinical, and psychological factors associated with digital and artificial intelligence literacy levels among both patient and control groups.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 50 years

Diagnosis of Fibromyalgia Syndrome according to 2016 American College of Rheumatology criteria (for patient group)

Adequate cognitive function

Literacy

Willingness to participate and provide informed consent

For control group: Healthy individuals matched by age and sex, with no reported health issues

Exclusion Criteria:

Cognitive impairment preventing questionnaire completion

Illiteracy

Presence of severe comorbidities or neurological/psychiatric disorders that may affect participation

Refusal or inability to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study included 106 patients diagnosed with Fibromyalgia Syndrome according to the 2016 American College of Rheumatology criteria and 106 age- and sex-matched healthy controls. Participants were aged between 18 and 50 years, literate, with adequate cognitive function, and voluntarily provided informed consent. The patient group was recruited from the Physical Medicine and Rehabilitation outpatient clinic at Yozgat Bozok University Faculty of Medicine. The control group consisted of healthy volunteers without any reported health issues.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
E-Health Literacy | At baseline"
  An 8-item, 5-point Likert-type scale developed by Norman and Skinner , validated in Turkish by Tamer Gencer. Higher scores indicate higher e- Health Literacy
Artificial Intelligence Literacy | At baseline"
  A 12-item, 7-point Likert-type scale developed by Wang et al . and adapted into Turkish by Çelebi et al . Higher scores indicate greater Artificial Intelligence literacy

SECONDARY OUTCOMES:
the Revised Fibromyalgia Impact Questionnaire | At baseline
  aims to measure patients with fibromyalgia syndrome status, progress and outcomes through 21 questions that inquire about physical functions, work-related situations, depression, anxiety, waking up tired, pain, stiffness, and fatigue The Turkish adaptation of the Revised Fibromyalgia Impact Questionnairewas psychometrically evaluated for validity and reliability by Sarmer et al .
the Beck Depression Inventory | At baseline
  is developed by Beck and colleagues in 1961, is intended to evaluate the typical signs and symptoms associated with depression. This instrument is a self-administered questionnaire comprising 21 items and usually requires around 10 minutes to complete. The Turkish version of the inventory was adapted and validated by Hisli and colleagues
Beck Anxiety Inventory | At baseline
  is developed by Aaron T. Beck, is an internationally validated tool for assessing anxiety levels. It consists of 21 items. The Turkish adaptation and validation of the inventory were performed by Ulusoy and colleagues

CONTACTS AND LOCATIONS:
Overall Officials: Gülseren Demir Karakılıç, Assistant Professor, Principal Investigator — Yozgat Bozok University
Locations (1):
- Yozgat Bozok University Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All data and materials are available upon reasonable requests from the corresponding author
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon study completion
Access Criteria: Researchers who provide a reasonable request and have a valid scientific purpose will be granted access to the individual participant data (IPD) and supporting documents, including the study protocol and informed consent form. Requests should be submitted to the corresponding author via email. Data sharing will be subject to approval to ensure participant confidentiality and compliance with ethical standards. Data will be shared in a de-identified format to protect participant privacy

REFERENCES:
- [Background] Çelebi, C., et al., Artificial intelligence literacy: An adaptation study. Instructional Technology and Lifelong Learning, 2023
- [Background] Wang, B., P.-L.P. Rau, and T. Yuan, Measuring user competence in using artificial intelligence: validity and reliability of artificial intelligence literacy scale. Behaviour & information technology, 2023
- [Background] TAMER GENCER, Z., Analysis of validity and reliability of Norman and Skinner's e-Health scale literacy for cultural adaptatio
- [Background] Norman CD, Skinner HA. eHealth Literacy: Essential Skills for Consumer Health in a Networked World. J Med Internet Res. 2006 Jun 16;8(2):e9. doi: 10.2196/jmir.8.2.e9. PMID 16867972
- [Background] Ulusoy, M., N.H. Sahin, and H. Erkmen, Turkish version of the Beck Anxiety Inventory: psychometric properties. Journal of cognitive psychotherapy, 1998
- [Background] Hisli, N., Beck depresyon envanterinin universite ogrencileri icin gecerliligi, guvenilirlig
- [Background] Sarmer S, Ergin S, Yavuzer G. The validity and reliability of the Turkish version of the Fibromyalgia Impact Questionnaire. Rheumatol Int. 2000 Dec;20(1):9-12. doi: 10.1007/s002960000077. PMID 11149662